CLINICAL TRIAL: NCT02660177
Title: Single Center, Open-label, Prospective Study to Characterize the Pharmacokinetics of Metamizole and Its Metabolites Following Intravenous Administration in Children Less Than 6 Years Old
Brief Title: Pharmacokinetics of Intravenous Metamizole in Children Less Than 6 Years Old
Acronym: PPMS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Children's Hospital Basel (Other)
Responsible Party: Principal Investigator, Frederique Rodieux, Dr. med, University Children's Hospital Basel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015-00020
Record Dates: First submitted 2016-01-14; First posted 2016-01-21 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Children; Pain; Surgery
MeSH Terms: conditions — Pain | interventions — Dipyrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- metamizole (Experimental): single IV metamizole (10mg/kg) administration
  Interventions: Drug: Metamizole

INTERVENTIONS:
Drug: Metamizole — metamizole IV administration
  Other Names: Novalgin

SUMMARY:
This study aims to assess the PK parameters of metamizole following a single IV administration of metamizole in children less than 6 years of age.

DETAILED DESCRIPTION:
This is an open-label pharmacokinetics (PK) study. It aims to assess the PK parameters of metamizole and its metabolites following a single IV administration of metamizole (10mg/kg) in children less than 6 years of age.

Thirty-nine children, 3-72 months of age, undergoing elective surgery at the University of Basel Children's Hospital, will receive, on the day of surgical procedure, a single dose of metamizole 10 mg/kg. After this dose, blood and saliva samples will be obtained at predetermined post-dose time points to measure concentrations of metamizole and its metabolites. The maximal duration of subject participation will be 24 hours. Plasma PK parameters (AUC, Cmax, Tmax, t1/2) of each analyte will be derived using noncompartmental methods. A population PK approach will be applied to characterize inter-subject variability and quantify the potential influence of age, sex and body weight on the PK parameters.

There are no published pharmacokinetic studies of metamizole in pediatrics. Furthermore, although Swissmedic provides no dose information for IV administration in infants with a body weight of less than 9 kg, IV is the most frequently used route of administration for direct postoperative analgesia in pediatrics, including infants with body weights of less than 9 kg. Due to the absence of data and the lack of any dosing recommendation for infants with a body weight less than 9 kg, the IV administration of metamizole in infants is "off-label" and inconsistent across hospitals and prescribing paediatricians.

ELIGIBILITY:
Inclusion Criteria:

* Infants and children 3-72 months of age at time of inclusion
* Body weight more than 5 kg at time of inclusion
* Children undergoing elective surgery at University of Basel Children's Hospital (UKBB) with planned administration of intravenous analgesia
* Patients who require surgical procedures that necessitate at least 24 hours in the hospital
* Parent/Legal guardian has been informed about the study and has signed Informed Consent Form

Exclusion Criteria:

* Infants and children who were born prematurely (before 37 weeks gestation), regardless of corrected gestational age
* Known kidney or liver disease
* Known neutropenia, anemia or other hematological disorders
* Known diagnosis of asthma
* Ongoing immunosuppression, except corticosteroid treatment, or primary immunodeficiency
* Treatment with strong inhibitors or inducers of CYP2C19 within 3 months prior to study
* Treatment with drugs known to induce agranulocytosis within 3 months prior to study
* Documented previous adverse reaction to metamizole
* Treatment with metamizole within 30 days prior to screening
* Any concomitant condition, which in the opinion of the investigator would preclude a subject's participation in the study
* Family members of investigators

Ages: 3 Months to 72 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2016-04; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curves (AUC0-inf, AUC0-24, AUC0-last) for metamizole and its metabolites in plasma and saliva | 0- 24 hours
  Time points of evaluation of these PK parameters: sampling at 1, 2, 4, 6, 10 and 24 hours after single IV metamizole dose.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) for metamizole and its metabolites in plasma and saliva | 0- 24 hours
  Time points of evaluation of these PK parameters: sampling at 1, 2, 4, 6, 10
Time to reach Cmax (tmax) for metamizole and its metabolites in plasma and saliva | 0- 24 hours
  Time points of evaluation of these PK parameters: sampling at 1, 2, 4, 6, 10
Terminal elimination rate constant with respective half-life time (t½) for metamizole and its metabolites in plasma and saliva | 0- 24 hours
  Time points of evaluation of these PK parameters: sampling at 1, 2, 4, 6, 10
Incidence of adverse events (AEs) | 0- 24 hours
Correlation between metamizole and its metabolites in saliva and plasma | 0- 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Marc Pfister, Professor, Principal Investigator — University Children's Hospital Basel; Rodieux Frederique, Dr. med, Principal Investigator — University Hospital, Geneva
Locations (1):
- UKBB, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ziesenitz VC, Rodieux F, Atkinson A, Borter C, Bielicki JA, Haschke M, Duthaler U, Bachmann F, Erb TO, Gurtler N, Holland-Cunz S, van den Anker JN, Gotta V, Pfister M. Dose evaluation of intravenous metamizole (dipyrone) in infants and children: a prospective population pharmacokinetic study. Eur J Clin Pharmacol. 2019 Nov;75(11):1491-1502. doi: 10.1007/s00228-019-02720-2. Epub 2019 Aug 7. PMID 31388703